CLINICAL TRIAL: NCT01489540
Title: Cost-effectiveness of Laser Doppler Imaging in Burn Care in the Netherlands
Brief Title: Cost-effectiveness of Laser Doppler Imaging in Burn Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association of Dutch Burn Centres (Other)
Collaborators: Dutch Burns Foundation (Other); Stichting Nuts Ohra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011-47
Record Dates: First submitted 2011-11-30; First posted 2011-12-09 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2011-12

CONDITIONS: Burns
Keywords: Burn; Depth; Diagnosis; Laser Doppler Imaging
MeSH Terms: conditions — Burns; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- new diagnostic strategy (Active Comparator): Combination of laser Doppler imaging and clinical assessment of burn depth
  Interventions: Device: laser Doppler imager (Moor)
- current diagnostic strategy (No Intervention): Clinical assessment of burn depth

INTERVENTIONS:
Device: laser Doppler imager (Moor) — The laser Doppler imager measures the blood flow of the skin/burn
  Other Names: Laser Doppler Imager, Moor Instruments; Moor LDI Burn Imager
  Arms: new diagnostic strategy

SUMMARY:
Accurate early burn depth assessment is important to determine the optimal treatment. The most applied method to asses burn depth is clinical assessment. This method is the least expensive, but not very accurate. Laser Doppler imaging (LDI) has been shown to accurately assess burn depth. The clinical effects, the costs and cost-effectiveness of this device however, are unknown. The hypothesis is that an eary accurate diagnosis will lead to an earlier therapeutic decision: surgery or no surgery. Earlier excision and grafting probably leads to a decrease in wound healing time, in length of hospital stay and in costs.

Before the investigators decide to implement LDI in Dutch burn care a study of the clinical effects and cost-effectiveness of LDI is necessary. Therefore a multicenter randomized controlled trial will be conducted, including all patients with burns of indeterminate depth (burns that are not obviously superficial or full thickness) treated in the Dutch burn centres. In total 200 patients will be included in an 18 months period. The patients are randomly divided in two groups: 'new diagnostic strategy' versus 'current diagnostic strategy'. Burn depth will be diagnosed both by clinical assessment and laser Doppler imaging in all patients. The results of the LDI-scan will be provided to the treating clinician in the 'new diagnostic strategy' group only. Time to wound healing, diagnostic and therapeutic decisions, and costs are observed.

ELIGIBILITY:
Inclusion criteria:

* Patients with acute burns of indeterminate depth (=intermediate depth, not obviously superficial or full thickness) at presentation
* Outpatient treatment or admission in one of the three Dutch burn centres
* Presentation within 5 days post burn

Exclusion criteria

* A presence of both burns of indeterminate depth and full thickness at presentation
* Patients with peri-orbital facial burns, in which the eyes are unable to shield
* Patients or their next of kin if they are under aged or temporary incompetent who can not be expected to give informed consent e.g. because of cognitive dysfunction or poor Dutch proficiency.
* Patients with a TBSA burned > 20%

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Wound healing time | 14 days post burn
  Time to complete wound healing (>95 % reepithelialisation) and rate of wound healing (% reepithelialisation) at day 14 post burn will be assessed clinically (Bloemen et al., 2011)

SECONDARY OUTCOMES:
The effect of LDI on patient outcomes: quality of life and scar quality | 3 months post burn
  Quality of life is measured with the EuroQol-5D in patient ≥ 5 years old (Bouillon et al., 2002) or the ItQol-47 in patients <5 years old (Raat et al., 2007):
  1. Baseline measurement within one month post burn
  2. Second measurement within 3 months post burn
  Scar quality is measured after 3 months:
  1. Scar elasticity with the Cutometer® Skin Elasticity Meter 575 (Draaijers et al., 2004)
  2. Vascularity and pigmentation with the Dermaspectometer (Draaijers et al., 2004)
  3. Self-reported scar quality: Patients Observer Scar Assessment Scale (van der Wal et al., 2011)
The effect of LDI on diagnostic and therapeutic decisions | Until wound healing, circa 2-6 weeks
  Effect of the introduction of the LDI will be assessed by comparing diagnostic decisions of burn clinicians, before and after the use of LDI.
  Possible diagnostic decisions are (Monstrey et al., 2011):
  * Superficial dermal burn, will heal (within 14 days)
  * Intermediate burn (possible will heal, or needs grafting)
  * Deep dermal or subdermal (full thickness) burn, needs grafting (will not heal within 21 days)
  The possible therapeutic decisions are:
  * Surgery
  * Postponement of decision
  * No surgery
The effect of LDI on total (medical and non medical) costs | From injury until 3 months post burn
  Costs from a societal perspective are calculated (following the Dutch guidelines from Oostenbrink et al., 2004):
  1. Costs during hospital stay
  2. Outpatient costs
  3. Non-hospital and non-medical costs
The cost-effectiveness of LDI compared to the standard diagnostic strategy | From injury until 3 months post burn
  In case of differences in patient outcome (wound healing time and scar quality) between both diagnostic strategies, cost-effectiveness will be calculated by dividing the difference in average costs by the difference in average time of wound healing or scar quality.
  In case of difference in quality of life between both diagnostic strategies, cost-utility will be calculated by dividing the difference in average costs by the difference in Quality Adjusted Life Years (QALY's).

CONTACTS AND LOCATIONS:
Overall Officials: Margriet E Baar, PhD, Study Chair — Associaton of Dutch Burns Centres
Locations (3):
- Netherlands (3):
  - Red Cross Hospital, Beverwijk, North Holland
  - Martini Hospital, Groningen, Provincie Groningen
  - Maasstad Hospital, Rotterdam, South Holland

REFERENCES:
- [Background] Kim LH, Ward D, Lam L, Holland AJ. The impact of laser Doppler imaging on time to grafting decisions in pediatric burns. J Burn Care Res. 2010 Mar-Apr;31(2):328-32. doi: 10.1097/BCR.0b013e3181d0f572. PMID 20182369
- [Background] Monstrey S, Hoeksema H, Verbelen J, Pirayesh A, Blondeel P. Assessment of burn depth and burn wound healing potential. Burns. 2008 Sep;34(6):761-9. doi: 10.1016/j.burns.2008.01.009. Epub 2008 Jun 3. PMID 18511202
- [Background] Jeng JC, Bridgeman A, Shivnan L, Thornton PM, Alam H, Clarke TJ, Jablonski KA, Jordan MH. Laser Doppler imaging determines need for excision and grafting in advance of clinical judgment: a prospective blinded trial. Burns. 2003 Nov;29(7):665-70. doi: 10.1016/s0305-4179(03)00078-0. PMID 14556723
- [Background] Engrav LH, Heimbach DM, Reus JL, Harnar TJ, Marvin JA. Early excision and grafting vs. nonoperative treatment of burns of indeterminant depth: a randomized prospective study. J Trauma. 1983 Nov;23(11):1001-4. doi: 10.1097/00005373-198311000-00007. PMID 6355500
- [Background] Herndon DN, Barrow RE, Rutan RL, Rutan TC, Desai MH, Abston S. A comparison of conservative versus early excision. Therapies in severely burned patients. Ann Surg. 1989 May;209(5):547-52; discussion 552-3. doi: 10.1097/00000658-198905000-00006. PMID 2650643
- [Background] Bloemen MC, van Zuijlen PP, Middelkoop E. Reliability of subjective wound assessment. Burns. 2011 Jun;37(4):566-71. doi: 10.1016/j.burns.2011.02.004. Epub 2011 Mar 8. PMID 21388743
- [Background] Bouillon B, Kreder HJ, Eypasch E, Holbrook TL, Kreder HJ, Mayou R, Nast-Kolb D, Pirente N, Schelling G, Tiling T, Yates D; MI Consensus Group. Quality of life in patients with multiple injuries--basic issues, assessment, and recommendations. Restor Neurol Neurosci. 2002;20(3-4):125-34. PMID 12454361
- [Background] Raat H, Landgraf JM, Oostenbrink R, Moll HA, Essink-Bot ML. Reliability and validity of the Infant and Toddler Quality of Life Questionnaire (ITQOL) in a general population and respiratory disease sample. Qual Life Res. 2007 Apr;16(3):445-60. doi: 10.1007/s11136-006-9134-8. Epub 2006 Nov 17. PMID 17111231
- [Background] Draaijers LJ, Botman YA, Tempelman FR, Kreis RW, Middelkoop E, van Zuijlen PP. Skin elasticity meter or subjective evaluation in scars: a reliability assessment. Burns. 2004 Mar;30(2):109-14. doi: 10.1016/j.burns.2003.09.003. PMID 15019116
- [Background] Draaijers LJ, Tempelman FR, Botman YA, Kreis RW, Middelkoop E, van Zuijlen PP. Colour evaluation in scars: tristimulus colorimeter, narrow-band simple reflectance meter or subjective evaluation? Burns. 2004 Mar;30(2):103-7. doi: 10.1016/j.burns.2003.09.029. PMID 15019115
- [Background] van der Wal MB, Tuinebreijer WE, Bloemen MC, Verhaegen PD, Middelkoop E, van Zuijlen PP. Rasch analysis of the Patient and Observer Scar Assessment Scale (POSAS) in burn scars. Qual Life Res. 2012 Feb;21(1):13-23. doi: 10.1007/s11136-011-9924-5. Epub 2011 May 20. PMID 21598065
- [Background] Monstrey SM, Hoeksema H, Baker RD, Jeng J, Spence RS, Wilson D, Pape SA. Burn wound healing time assessed by laser Doppler imaging. Part 2: validation of a dedicated colour code for image interpretation. Burns. 2011 Mar;37(2):249-56. doi: 10.1016/j.burns.2010.08.013. Epub 2010 Nov 16. PMID 21084164
- [Derived] Hop MJ, Stekelenburg CM, Hiddingh J, Kuipers HC, Middelkoop E, Nieuwenhuis MK, Polinder S, van Baar ME; LDI Study Group. Cost-Effectiveness of Laser Doppler Imaging in Burn Care in The Netherlands: A Randomized Controlled Trial. Plast Reconstr Surg. 2016 Jan;137(1):166e-176e. doi: 10.1097/PRS.0000000000001900. PMID 26710049
- [Derived] Hop MJ, Hiddingh J, Stekelenburg C, Kuipers HC, Middelkoop E, Nieuwenhuis MK, Polinder S, van Baar ME; LDI study group. Cost-effectiveness of laser Doppler imaging in burn care in the Netherlands. BMC Surg. 2013 Feb 1;13:2. doi: 10.1186/1471-2482-13-2. PMID 23369360